CLINICAL TRIAL: NCT06647615
Title: A Pilot Study to Assess the Safety, Tolerability, and Efficacy of Virtual Reality for the Treatment of Abdominal Pain in Quiescent Crohn's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jami A. Kinnucan, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-001863
Record Dates: First submitted 2024-10-15; First posted 2024-10-18 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Crohn's Disease; Abdominal Pain (AP)
Keywords: Crohn's Disease; Quiescent Crohn's Disease
MeSH Terms: conditions — Crohn Disease; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- VR Headset (Experimental)
  Interventions: Device: VR headset

INTERVENTIONS:
Device: VR headset — The VR portion of the study will last for 8 weeks. You will be asked to use your headset on a daily basis for at least 30 minutes, but you are free to use the headset as much as you would like.

SUMMARY:
The purpose of this research is to see if patients with Crohn's disease (CD) and abdominal pain resulting in health-related quality of life deficits despite lack of evidence of active inflammation improve with the use of virtual reality (VR).

DETAILED DESCRIPTION:
The goal of this research is to see if patients with Crohn's disease (CD) and abdominal pain resulting in health-related quality of life deficits despite lack of evidence of active inflammation improve with the use of virtual reality (VR). The use of VR therapy is investigational. You have been asked to take part in this research because you have been identified as an adult with CD with abdominal pain at least weekly despite normal C-reactive protein and fecal calprotectin levels in adult patients, age 18- 70 years old. Demographic information will be gathered (age, sex, race, current medication use, co-morbid conditions), as will prior tests and interventions.

Participants will be asked to participate in the two-week pre-screening evaluation for symptoms through questionnaires. The VR portion of the study will last for 8 weeks. You will be asked to use your headset on a daily basis for at least 30 minutes, but you are free to use the headset as much as you would like. You will be called on a weekly basis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of endoscopically and histologically confirmed CD with evidence of C-reactive protein < 5 mg/dL and fecal calprotectin < 150microg/g who also report any abdominal pain at least weekly will be included.

Exclusion Criteria:

* Patients will be excluded from the study if they do not have biopsy-proven CD, have a known seizure disorder, if symptoms are thought to represent an organic disorder, those with visual or hearing impairments, if symptoms represent a known pelvic floor disorder, if the patient is using opioids, has significant ongoing psychological distress (HAD score > 11 for either anxiety or depression), or if the patient can not actively participate in the study for any other reason (e.g., inability to understand English as the VR program as an English only).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in abdominal pain | 10 weeks
  Improvement in mean abdominal pain by 25% at week 10 as compared to baseline in patients with quiescent CD using the 0-10 Likert pain scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kinnucan, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Furlan AD, Sandoval JA, Mailis-Gagnon A, Tunks E. Opioids for chronic noncancer pain: a meta-analysis of effectiveness and side effects. CMAJ. 2006 May 23;174(11):1589-94. doi: 10.1503/cmaj.051528. PMID 16717269
- [Background] Noureldin M, Higgins PDR, Govani SM, Cohen-Mekelburg S, Kenney BC, Stidham RW, Waljee JF, Waljee AK. Incidence and predictors of new persistent opioid use following inflammatory bowel disease flares treated with oral corticosteroids. Aliment Pharmacol Ther. 2019 Jan;49(1):74-83. doi: 10.1111/apt.15023. Epub 2018 Nov 14. PMID 30430615
- [Background] Wiederhold BK, Gao K, Sulea C, Wiederhold MD. Virtual reality as a distraction technique in chronic pain patients. Cyberpsychol Behav Soc Netw. 2014 Jun;17(6):346-52. doi: 10.1089/cyber.2014.0207. PMID 24892196
- [Background] Tashjian VC, Mosadeghi S, Howard AR, Lopez M, Dupuy T, Reid M, Martinez B, Ahmed S, Dailey F, Robbins K, Rosen B, Fuller G, Danovitch I, IsHak W, Spiegel B. Virtual Reality for Management of Pain in Hospitalized Patients: Results of a Controlled Trial. JMIR Ment Health. 2017 Mar 29;4(1):e9. doi: 10.2196/mental.7387. PMID 28356241
- [Background] Lacy BE, Cangemi DJ, Spiegel BR. Virtual Reality: A New Treatment Paradigm for Disorders of Gut-Brain Interaction? Gastroenterol Hepatol (N Y). 2023 Feb;19(2):86-94. PMID 36866110
- [Background] Docherty MJ, Jones RC 3rd, Wallace MS. Managing pain in inflammatory bowel disease. Gastroenterol Hepatol (N Y). 2011 Sep;7(9):592-601. PMID 22298998